CLINICAL TRIAL: NCT03476642
Title: A Volunteer Study to Determine the Anatomical Distribution of Injectate, the Extent of Sensory Block, and the Pharmacokinetics of Ropivacaine Following Erector Spinae Plane (ESP) Blocks.
Brief Title: Distribution, Pharmacokinetics and Extent of Sensory Blockade in ESP Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sanjib D Adhikary, Associate Professor, Director Acute Pain, Regional Anesthesia/Ortho, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY0008641
Record Dates: First submitted 2018-03-01; First posted 2018-03-26 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Distribution of Ropivacaine in Erector Spinae Plane Block
MeSH Terms: interventions — Ropivacaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: This will be a randomized,double blinded, controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine with Epinephrine (Active Comparator): Group RE will have 20mL of 0.5% Ropivacaine with epinephrine injected at the left or right T5 transverse process.
  Interventions: Drug: Ropivacaine; Drug: Epinephrine
- Ropivacaine without Epinephrine (Active Comparator): Group R will have 20mL of 0.5% Ropivacaine without epinephrine injected at the left or right T5 transverse process.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — injection of 20mL of 0.5% Ropivacaine at the left or right T5 transverse process
Drug: Epinephrine — injection of 20mL epinephrine in combination with ropivacaine at the left or right T5 transverse process
  Arms: Ropivacaine with Epinephrine

SUMMARY:
The primary objectives of this study are to define the extent of dermatomal anesthesia and anatomical spread of injectate (as defined by MRI imaging) that is provided by an ESP block at the T5 level, using twenty milliliters of 0.5% ropivacaine.

The secondary objectives include: 1) the measurement of changes in hemodynamic parameters associated with the ESP block, 2) the duration of sensory effects provided by ropivacaine with or without epinephrine, 3) the venous plasma concentration of ropivacaine associated at various time intervals after completion of the ESP block.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 60 inclusive
* Weight between 60 and 100 kg inclusive
* Height 160 to190 cm inclusive

Exclusion Criteria:

* Pregnant females
* Chronic medical condition requiring medication
* History of previous major spinal, abdominal or thoracic surgery
* Congenital abnormalities of the spine, back, thorax or abdomen
* History of major trauma to the thorax or abdomen;
* Allergy to ropivacaine or other amide local anesthetics
* The presence of any metallic implant in their body
* Any contraindication to magnetic resonance imaging as determined by completion of a standard questionnaire administered to all patients undergoing magnetic resonance imaging.
* Allergy to Gadolinium radiological contrast agent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjib Adhikary, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S.Hershey Medical center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.5% Ropivacaine With Epinephrine: no adverse events
- 0.5% Ropivacaine Without Epinephrine: No advere events
Period: Overall Study
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 0.5% Ropivacaine With Epinephrine: 20mL of 0.5% Ropivacaine with epinephrine injected at the left or right T5 transverse process.
- 0.5% Ropivacaine Without Epinephrine: 0.5% Ropivacaine without epinephrine injected at the left or right T5 transverse process.
- Total: Total of all reporting groups
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 42 [25 to 59] | 31 [23 to 54] | 37 [23 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Area of Dermatomal Sensory Loss at 20 Min
Description: A consultant anesthesiologist blinded to the randomization allocation will perform a sensory assessment for loss of sensation to cold using ethanol on the skin
Time Frame: 20 minutes from the time of the ESP block
Measure: Mean (Standard Deviation); unit: cm^2
Groups:
- 0.5% Ropivacaine Without Epinephrine: 20mL of 0.5% Ropivacaine without epinephrine injected at the left or right T5 transverse process.
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Number analyzed (Participants) | 6 | 6
cm^2 | 68.8 (43.7) | 167.5 (178.0)

2. Primary Outcome: Area of Dermatomal Sensory Loss 60 Min
Description: as for outcome 1
Time Frame: 60 minutes from the time of the ESP block
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Number analyzed (Participants) | 6 | 6
cm^2 | 90.2 (43.9) | 61.0 (37.1)

3. Primary Outcome: Area of Dermatomal Sensory Loss 120 Min
Description: as for outcome 1
Time Frame: 120 minutes from the time of the ESP block
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Number analyzed (Participants) | 6 | 6
cm^2 | 107.1 (69.8) | 109.1 (125.0)

4. Primary Outcome: Area of Dermatomal Sensory Loss at 240 Min
Description: as for outcome 1
Time Frame: 240 minutes from the time of the ESP block
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Number analyzed (Participants) | 6 | 6
cm^2 | 55.5 (36.0) | 114.5 (170.8)

5. Primary Outcome: Area of Dermatomal Sensory Loss 360 Min
Description: as for outcome 1
Time Frame: 360 minutes from the time of the ESP block
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Number analyzed (Participants) | 6 | 6
cm^2 | 35.0 (46.1) | 12.9 (24.3)

6. Primary Outcome: Venous Plasma Concentration of Ropivacaine at 20 Min
Description: 3 ml of blood will be obtained from the Intravenous line already placed in the subject prior to performing the block.
Time Frame: These samples will be repeated at 20 minutes after completion of the injection of active drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Number analyzed (Participants) | 6 | 6
ng/mL | 599.6 (187.2) | 1284.7 (336.5)

7. Primary Outcome: Venous Plasma Concentration of Ropivacaine at 60 Min
Description: 3 ml of blood will be obtained from the Intravenous line already placed in the subject prior to performing the block.
Time Frame: These samples will be repeated at 60 minutes after completion of the injection of active drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Number analyzed (Participants) | 6 | 6
ng/mL | 669.0 (114.4) | 962.4 (365.3)

8. Primary Outcome: Venous Plasma Concentration of Ropivacaine at 90 Min
Description: 3 ml of blood will be obtained from the Intravenous line already placed in the subject prior to performing the block.
Time Frame: These samples will be repeated at 90 minutes after completion of the injection of active drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Number analyzed (Participants) | 6 | 6
ng/mL | 625.9 (171.9) | 837.9 (349.3)

9. Primary Outcome: Venous Plasma Concentration of Ropivacaine at 120 Min
Description: 3 ml of blood will be obtained from the Intravenous line already placed in the subject prior to performing the block.
Time Frame: These samples will be repeated at 120 after completion of the injection of active drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Number analyzed (Participants) | 6 | 6
ng/mL | 640.0 (129.5) | 691.6 (289.9)

10. Primary Outcome: Venous Plasma Concentration of Ropivacaine at 240 Min
Description: 3 ml of blood will be obtained from the Intravenous line already placed in the subject prior to performing the block.
Time Frame: These samples will be repeated at 240 minutes after completion of the injection of active drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Number analyzed (Participants) | 6 | 6
ng/mL | 480.3 (99.0) | 420.9 (183.5)

11. Primary Outcome: Volume of Injectate Spread Measured Using MRI at 30 Min
Description: The subject will undergo two MRIs to determine the spread of the anesthetic.
Time Frame: 30 minutes from the time of the ESP block
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Number analyzed (Participants) | 6 | 6
mm^3 | 4373.2 (1013.5) | 3712.8 (1011.3)

12. Primary Outcome: Volume of Injectate Spread Measured Using MRI at 90 Min
Description: The subject will undergo two MRIs to determine the spread of the anesthetic.
Time Frame: 90 minutes from the time of the ESP block
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | 0.5% Ropivacaine With Epinephrine | 0.5% Ropivacaine Without Epinephrine
Number analyzed (Participants) | 6 | 6
mm^3 | 3863.0 (944.6) | 3751.2 (1197.2)

ADVERSE EVENTS:
Time Frame: up to 48 hour following intervention
Groups:
- Group With EPI: No adverse Effects for the study
- Group Without Epi: No adverse events
Arm/Group | Group With EPI | Group Without Epi
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/42/NCT03476642/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT03476642/ICF_001.pdf